CLINICAL TRIAL: NCT07057700
Title: Investigating the Mechanisms of Welwalk Robot in Restoring Motor Function of the Lower Extremities in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing Xie, PhD, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025230
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Walking Impairment
Keywords: stroke; Lower limb dysfunction; robotics; gait
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- welwalk training (Experimental): Daily physiotherapy training using the welwalk lower limb walking training robot
  Interventions: Device: welwalk training
- conventional physical therapy (Active Comparator): Daily training using traditional physiotherapy such as core training, gait training, etc.
  Interventions: Other: physical therapy

INTERVENTIONS:
Device: welwalk training — welwalk training group 30 min of welwalk robot-assisted training + 15 min of walking training + 15 min of other training per session.The intervention lasted a total of 3 weeks, 6 sessions/week, 1 hour/session.
  Arms: welwalk training
Other: physical therapy — 45 min of walking training + 15 min of other training per session. The intervention lasted a total of 3 weeks, 6 sessions/week, 1 hour/session.
  Arms: conventional physical therapy

SUMMARY:
Current evidence and clinical applications of robotic gait training devices for motor function recovery post-stroke are increasingly available. Although existing research demonstrates that robotic gait training can improve patients' gait and balance, there remains a lack of in-depth investigation into its specific mechanisms of action concerning central nervous system (CNS) reorganization - notably, changes in activity within the motor cortex and associated neural networks. The intrinsic changes within the CNS have received insufficient attention, limiting a comprehensive and profound understanding of the rehabilitation outcomes. Therefore, this study aims to elucidate the potential mechanisms underlying robotic gait training-induced neuroplasticity by integrating functional near-infrared spectroscopy (fNIRS) technology with multi-dimensional lower limb motor function assessment tools (such as FAC, BBS, AMEDA, 10MWT, 6MWT, TUGT). It will systematically investigate the effects of robotic gait training on both the central nervous system and lower limb motor function in stroke patients. Furthermore, the study will compare the differences in functional recovery efficacy between robotic gait training and conventional rehabilitation therapies.

DETAILED DESCRIPTION:
In this study, participants will be randomly allocated into two groups: the Welwalk training group and the conventional rehabilitation therapy group.

Welwalk Training Group: Each session will consist of 30 minutes of Welwalk robot-assisted training, followed by 15 minutes of gait training and 15 minutes of supplementary exercises.Control Group (Conventional Rehabilitation Therapy): Each session will consist of 45 minutes of gait training and 15 minutes of supplementary exercises.The intervention period will span 3 weeks, with sessions administered six times per week. Each session will last 1 hour.

Clinical assessments will be conducted by certified healthcare professionals at four time points: at baseline (prior to the commencement of formal training), and after the 1st week, 2nd week, and 3rd week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients or family gave written informed consents to participate in this study.
* Patients with first hemiplegia caused by primary supratentorial intracerebral hemorrhage or cerebral infarction.
* Within 1 year of stroke onset
* Aged ≥ 20
* Body weight is between 40 and 80 kg
* No excessive spasticity in hip, knee, and ankle joints (Modified Ashworth Scale <3)
* sufficient cognition to follow simple instructions and to understand the content and purpose of the study (Chinese version-MOCA ≥ 20 points)
* Patients who have risks of giving-way when they walk with Ankle-Foot orthosis (AFO)

Exclusion Criteria:

* A history of myocardial infarction
* Muscular or neurological disorder including diabetic neuropathy
* Symptomatic angina or arrhythmia
* Symptomatic respiratory disorder
* Communicable infection
* Joint contracture or limb deformity that affects walking (Range of motion of hip extension < 5 degree, knee extension < -5 degree (can be flexible), ankle dorsiflexion with knee extension position < 5 degree)
* Heterotropic ossification that restrict the range of motion of joints of lower extremities
* Being vulnerable to fracture like severe osteoporosis of spine or lower extremities
* Incontinence of urine or feces that may deface the robotic knee-ankle-foot device of Welwalk
* Inadequate control of hypertension (resting systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 120 mmHg)
* Inadequate control of tachycardia (heart rate at rest ≥ 120 bpm)
* Training restriction due to reduced cardiac function or respiratory dysfunction
* Visual or auditory impairment hindering training
* Pregnant patients
* Recent participation in other clinical trials
* Patient whom examination doctor judge improper as a trial subject
* Anyone not able to sustain the training protocol with Welwork or regular training

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The Functional Ambulation Categories (FAC) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3);
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.The FAC uses a six-point scale from 0 to 5, where a higher score indicates better performance.

SECONDARY OUTCOMES:
functional near - infrared spectroscopy (fNIRS) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  Using fNIRS technology to observe brain activation and brain network changes during the walking period in participants.
10 Meter Walk Test(10WMT) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  assessing the participants' walking ability. Less time spent by patients indicates better walking ability.
Timed Up and Go Test (TUGT) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  Assessment of motor function of the unaffeected and affected steering sides
6minute walking test(6MWT) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  Assessment of cardiorespiratory endurance in participants
Berg Balance Scale (BBS) | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  Assessment of the participant's ability to balance. The BBS is scored on a scale of 0 to 56; higher scores reflect better balance function.
Modified Barthel Index,MBI | Before intervention (Week 0); After the First week of intervention (Week 1); After the Second week of intervention (Week 2); After the Third week of intervention (Week 3)
  Assessment of the subject's ability to perform daily living tasks.The MBI is scored on a scale of 0 to 100; higher scores reflect better ADL.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, affiliated to Shanghai Jiao Tong University, School of medicine,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the demographic information and baseline clinical data of all participants.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Authorized professional researchers, including but not limited to researchers engaged in neuroscience research who have obtained data access permission from their affiliated institutions, and clinical doctors from other medical institutions that have a cooperative relationship with this study and have signed data confidentiality agreements.
  They can access the detailed clinical medical histories of the participants, including past disease histories and treatment process records; neurological function assessment scale data; as well as imaging data collected during the study, such as brain magnetic resonance imaging (MRI) results. However, sensitive information related to participants' privacy, such as names, ID numbers, and contact information, will be strictly anonymized to ensure that such information cannot be obtained.
  They can contact the corresponding author or the first author via email.

REFERENCES:
- [Background] Zhang B, Li D, Liu Y, Wang J, Xiao Q. Virtual reality for limb motor function, balance, gait, cognition and daily function of stroke patients: A systematic review and meta-analysis. J Adv Nurs. 2021 Aug;77(8):3255-3273. doi: 10.1111/jan.14800. Epub 2021 Mar 6. PMID 33675076
- [Background] Wang C, Zhang Q, Hou S, Guo D, Han X, Huo W, Zhang Y. Split-belt treadmill training improves gait symmetry and lower limb function in patients with stroke. Sci Rep. 2025 May 8;15(1):16123. doi: 10.1038/s41598-025-98322-3. PMID 40341197
- [Background] Sheng Y, Han J. Biomechanical characteristics and neuromuscular action control mechanism of single-dual-task walking-conversion training in stroke patients. J Back Musculoskelet Rehabil. 2025 May;38(3):576-592. doi: 10.1177/10538127241308215. Epub 2025 Feb 12. PMID 39973293
- [Background] Caliandro P, Molteni F, Simbolotti C, Guanziroli E, Iacovelli C, Reale G, Giovannini S, Padua L. Exoskeleton-assisted gait in chronic stroke: An EMG and functional near-infrared spectroscopy study of muscle activation patterns and prefrontal cortex activity. Clin Neurophysiol. 2020 Aug;131(8):1775-1781. doi: 10.1016/j.clinph.2020.04.158. Epub 2020 May 18. PMID 32506008
- [Background] Li X, Zhang H, Zhang W, Wu J, Dai L, Long N, Jin T, Gu L, Chen J. Neural mechanisms underlying the improvement of gait disturbances in stroke patients through robot-assisted gait training based on QEEG and fNIRS: a randomized controlled study. J Neuroeng Rehabil. 2025 Jun 18;22(1):136. doi: 10.1186/s12984-025-01656-2. PMID 40533805
- [Background] Belda-Lois JM, Mena-del Horno S, Bermejo-Bosch I, Moreno JC, Pons JL, Farina D, Iosa M, Molinari M, Tamburella F, Ramos A, Caria A, Solis-Escalante T, Brunner C, Rea M. Rehabilitation of gait after stroke: a review towards a top-down approach. J Neuroeng Rehabil. 2011 Dec 13;8:66. doi: 10.1186/1743-0003-8-66. PMID 22165907
- [Background] Fan T, Zheng P, Zhang X, Gong Z, Shi Y, Wei M, Zhou J, He L, Li S, Zeng Q, Lu P, Zhao Y, Zou J, Chen R, Peng Z, Xu C, Cao P, Huang G. Effects of exoskeleton rehabilitation robot training on neuroplasticity and lower limb motor function in patients with stroke. BMC Neurol. 2025 May 3;25(1):193. doi: 10.1186/s12883-025-04203-7. PMID 40319228
- [Background] Chen S, Zhang W, Wang D, Chen Z. How robot-assisted gait training affects gait ability, balance and kinematic parameters after stroke: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2024 Jun;60(3):400-411. doi: 10.23736/S1973-9087.24.08354-0. Epub 2024 Apr 22. PMID 38647534
- [Background] Hao QH, Qiu MM, Wang J, Tu Y, Lv ZH, Zhu TM. The effect of lower limb rehabilitation robot on lower limb -motor function in stroke patients: a systematic review and meta-analysis. Syst Rev. 2025 Mar 26;14(1):70. doi: 10.1186/s13643-025-02759-6. PMID 40140968
- [Background] Zhang S, Fan L, Ye J, Chen G, Fu C, Leng Y. An Intelligent Rehabilitation Assessment Method for Stroke Patients Based on Lower Limb Exoskeleton Robot. IEEE Trans Neural Syst Rehabil Eng. 2023;31:3106-3117. doi: 10.1109/TNSRE.2023.3298670. Epub 2023 Aug 2. PMID 37490379
- [Background] Hesse S, Mehrholz J, Werner C. Robot-assisted upper and lower limb rehabilitation after stroke: walking and arm/hand function. Dtsch Arztebl Int. 2008 May;105(18):330-6. doi: 10.3238/arztebl.2008.0330. Epub 2008 May 2. PMID 19629252
- [Background] Xu S, Zhu S, Li M, Zhang T, Wang Q, Sui Y, Shen Y, Chaojie K, Zhuang R, Guo C, Wang T, Zhu L. Altered cortical activation patterns in post-stroke patients during walking with two-channel functional electrical stimulation: a functional near-infrared spectroscopy observational study. Front Neurol. 2025 Jan 13;15:1449667. doi: 10.3389/fneur.2024.1449667. eCollection 2024. PMID 39871991
- [Background] Rodriguez-Fernandez A, Lobo-Prat J, Font-Llagunes JM. Systematic review on wearable lower-limb exoskeletons for gait training in neuromuscular impairments. J Neuroeng Rehabil. 2021 Feb 1;18(1):22. doi: 10.1186/s12984-021-00815-5. PMID 33526065
- [Background] Scrivener K, Dorsch S, McCluskey A, Schurr K, Graham PL, Cao Z, Shepherd R, Tyson S. Bobath therapy is inferior to task-specific training and not superior to other interventions in improving lower limb activities after stroke: a systematic review. J Physiother. 2020 Oct;66(4):225-235. doi: 10.1016/j.jphys.2020.09.008. Epub 2020 Oct 14. PMID 33069609